CLINICAL TRIAL: NCT04299750
Title: Impact of Alveolar Ridge Preservation on Optimal Implant Placement
Brief Title: Impact of a Alveolar Ridge Preservation Technique on the Need of Performing Guided Bone Regeneration for Dental Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Simone Lumetti (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry); Geistlich Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Simone Lumetti, DDS, PhD, MSc, University of Parma
Organization: University of Parma (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sockpres-13
Record Dates: First submitted 2015-05-03; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Tooth Avulsion
Keywords: Socket preservation; Single implant; Tooth extraction
MeSH Terms: conditions — Tooth Avulsion | interventions — Tooth Extraction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Alveolar Ridge Preservation (Experimental): Patients in this arm will undergo atraumatic extraction of an hopeless tooth and a socket preservation procedure. Alveolar ridge preservation will be performed using a slow-resorption bone substitute and a collagen membrane that covers the graft.
  Interventions: Procedure: Tooth extraction and Alveolar ridge preservation
- Natural healing (Active Comparator): Patients in this arm will undergo atraumatic extraction of an hopeless tooth. The socket will follow natural healing.
  Interventions: Procedure: Tooth extraction

INTERVENTIONS:
Procedure: Tooth extraction and Alveolar ridge preservation — Tooth extraction and alveolar ridge preservation with deproteinized bovine bone mineral and a collagen matrix seal
  Other Names: Socket preservation
  Arms: Alveolar Ridge Preservation
Procedure: Tooth extraction — Tooth extraction and socket natural healing
  Other Names: Socket natural healing
  Arms: Natural healing

SUMMARY:
The aim of this study is to investigate how a socket preservation procedure may reduce the need of guided bone regeneration surgery after tooth extraction and facilitate the placement of a dental implant in the optimal, prosthetic-driven position.

DETAILED DESCRIPTION:
The main gol of the study is to assess the efficacy of a socket preservation procedure in reducing the need of additional surgeries in order to augment alveolar bone volume before placing a dental implant in optimal position. Bone volume at 6 months will be compared to initial volume in order to assess volume variations and how they affect the positioning of a prosthetically driven, implant.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age

  * at least one intercalate tooth to be extracted, with complete alveolus and no soft tissue recession;
  * adequate oral hygiene, i.e. plaque index score ≤10%;
  * mesial-distal width of inter-dental space ≥7 mm;

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) score ≥III
* presence of active periodontitis, clinically diagnosed in presence of probing depths ≥4 mm and bleeding on probing
* a history of radiotherapy to the head and neck region
* presence of conditions requiring chronic use of antibiotics
* medical conditions requiring prolonged use of steroids
* history of leucocyte dysfunction
* history of bleeding disorders
* history of renal failure
* patients with metabolic bone disorders
* patients with uncontrolled endocrine disorders
* disability affecting oral hygiene
* alcohol or drug abuse
* HIV infection
* smoking >10 cigarettes a day or cigar equivalents
* conditions or circumstances that would prevent completion of study participation
* mucosal diseases
* presence of osseous lesions
* severe bruxing or clenching habits
* persistent intraoral infections
* compromised alveolus (dehiscence, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Number of implants ideally placed | 6 months
  The main goal is to determine if alveolar ridge preservation affects optimal implant positioning. This is defined as the implant position allowing to fulfill the ideal prosthetic design of the crown to be restored.

SECONDARY OUTCOMES:
Peri-implant bone variation | 6 months
  Crestal bone levels (CBL): distances from the implant shoulder to the most coronal bone to implant contact measured on X-rays with a millimeter ruler to the nearest 0.5 mm. Two measurements will be taken for each implant: mesially and distally
Ridge volume at 6 months after tooth extraction | 6 months
  The comparison of baseline and control cone.beam computed tomography and of clinical data in test and control groups will allow to determine volumetric effects on bone and soft tissues of socket preservation.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Macaluso, MDS, MSc, Study Director — University of Parma
Locations (1):
- Centro Universitario di Odontoiatria, Parma, PR, Italy